CLINICAL TRIAL: NCT05522946
Title: Circle Game Collaborative--Freddie the Frog
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants were not assigned to an intervention and as such this was not considered a clinical trial.
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020B0306
Record Dates: First submitted 2021-04-01; First posted 2022-08-31 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Impairment; Physical Disability
Keywords: Children with disabilities; Parent; Family; Games; Technology; Collaborative game
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Group 1: Parents and children without disabilities Group 2: Parents and adolescents with mild to moderate cognitive or physical disability Group 3: Parents and adolescents with moderate to severe cognitive and/or physical disability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parent and child without disability (Experimental): Parent and child will play the game on the iPad using the sensors provided.
  Interventions: Other: Gameplay between parent and child or adolescent with or without a disability
- Parent and adolescent with mild to moderate cognitive or physical disability (Experimental): Parent and adolescent will play the game on the iPad using the sensors provided.
  Interventions: Other: Gameplay between parent and child or adolescent with or without a disability
- Parent and adolescent with moderate to severe cognitive and/or physical disability (Experimental): Parent and adolescent will play the game on the iPad using the sensors provided.
  Interventions: Other: Gameplay between parent and child or adolescent with or without a disability

INTERVENTIONS:
Other: Gameplay between parent and child or adolescent with or without a disability — Parent and child or adolescent will play the game using the provided sensors for 10-15 minutes total. Depending on the cognitive and/or physical ability of the child or adolescent, the two may take turns wearing the sensors or if the child or adolescent does not have the physical or cognitive ability to deliberately touch the sensor, then the child or adolescent will wear the sensors and the parent will touch the sensors in order to move the game forward.

SUMMARY:
Families who have children with disabilities experience more challenges in interacting with their children than families who have children without disabilities. This increased level of burden results in higher rates of emotional stress and hardship for those families. Motivated by the idea of making deeper connections between children with disabilities and their parents, our gaming platform is designed around two key concepts - human touch and collaborative play. Using wearable sensors, conductive fabrics, microcontrollers, and wireless communication, our gaming platform will register and interpret "touch" as a way to interface with game apps and the devices they are installed on. In other words, touch is translated into player input. Thus, rather than interact with an iPad directly, children and their parents interact with each other instead. Our platform engages both parents and children with disabilities equally in order to better focus on their shared physical expression. As touch can be registered from any part of the body, our platform can be used with children with any type of disability and allows for both active and passive participation by children with a severe disability.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Children without disabilities between the ages of 5-9 years. Any parent/caregiver to the child

Group 2: Adolescents with mild to moderate physical or cognitive disability between the ages of 10-17 years. Any parent/caregiver to the child

Group 3: Adolescents with moderate to severe physical and/or cognitive disability between the ages of 10-17 years. Any parent/caregiver to the child

Exclusion Criteria:

All groups:

* Parents who do not understand and speak English
* Parents with a disability

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Establish the feasibility of cooperative gameplay between parents and children without disabilities | 1 hour
  Successful completion of gameplay session
Establish the feasibility of cooperative gameplay between parents and adolescents with disabilities | 1 hour
  Successful completion of gameplay session
Examine childs', adolescents', and parents ability to play the game through analysis of video recordings of game play | 1 hour
  Successful completion of gameplay session

SECONDARY OUTCOMES:
Explore childs' and adolescents' Global, Mental, Physical, and Social Health using the Patient-Reported Outcomes Measurement Information System (PROMIS) measure | Pre-gameplay
  Using individual Patient-Reported Outcomes Measurement Information System (PROMIS) items from the global health, mental health, physical health, social health, and symptom item banks, explore the child and adolescent global health, mental health, physical health, social health, as well as pain and stress. The scores will range from 2-54 with higher scores indicating better outcomes.
Semi-Structured interviews with open-ended questions to explore childs' and adolescents' (where appropriate), and parents' feelings about gameplay for fun, well being, quality of life | Immediately Post-gameplay and up to one week post-gameplay
  Using semi-structured interviews with open ended questions, we will ask parents and children/adolescents who are willing and able to answer questions related to playing the game together. We will ask children/adolescents who are willing and able questions immediately post gameplay. We will ask parents questions related to gameplay either immediately after the child/adolescent or up to 1 week later. To be qualitatively analyzed
Explore the parents' feelings of bonding with their child/adolescent using the "Connection & Bonding Questionnaire" | 1 hour post-game play
  Explore parent feelings of bonding pre/post gameplay examine whether playing the game together increased their feelings of bonding with their child/adolescent. Bonding will be measured using a new investigator-developed measure named the Connection & Bonding Questionnaire, a 5 item Likert-style questionnaire with responses ranging from Strongly Disagree (0) to Strongly Agree (5) and scores ranging from 0-25 with higher scores indicating a stronger connection and parent/child bond.
Explore whether the parent felt that their child's physical and psychological needs were met before gameplay using the "Child Needs Survey" | Pre-gameplay
  Explore whether the parent felt that their child's physical and psychological needs were met before gameplay using an investigator-developed measure named the "Child Needs Survey", a 5 item survey with 4 questions with responses of Yes, No, Unsure/Decline to Answer, and Not able/Not applicable, one visual analog-type response ranging from "Little to none" to "Fully" and one open-ended question asking parents to describe any additional needs that may or may not have been met. More "yes" answers mean a better outcome.
Explore whether the child had pain pre/post gameplay using visual analog scale | Pre gameplay and immediately post gameplay
  Using a visual analog scale, have the child and parent rate the child's pain pre- and immediately post-gameplay. Visual Analog Scales are a 100mm line with endpoints "none" at the 0 endpoint and "worst ever" at the 100mm endpoint. A higher score indicates a worse outcome.
Explore whether the child had stress pre/post gameplay using visual analog scale | Pre gameplay and immediately post gameplay
  Using a visual analog scale, have the child and parent rate the child's stress pre- and immediately post-gameplay. Visual Analog Scales are a 100mm line with endpoints "none" at the 0 endpoint and "worst ever" at the 100mm endpoint. A higher score indicates a worse outcome.
Explore whether the parent had pain pre/post gameplay using visual analog scale | Pre gameplay and immediately post gameplay
  Using a visual analog scale, have the parent rate their pain pre- and immediately post-gameplay. Visual Analog Scales are a 100mm line with endpoints "none" at the 0 endpoint and "worst ever" at the 100mm endpoint. A higher score indicates a worse outcome.
Explore whether the parent had stress pre/post gameplay using visual analog scale | Pre gameplay and immediately post gameplay
  Using a visual analog scale, have the parent rate the their stress pre and immediately post gameplay. Visual Analog Scales are a 100mm line with endpoints "none" at the 0 endpoint and "worst ever" at the 100mm endpoint. A higher score indicates a worse outcome.
Compare childs' and adolescents' Global, Mental, Physical, and Social Health using the single measure "Patient-Reported Outcomes Measurement Information System (PROMIS)" from Group 1, Group 2, and Group 3 | 1 hour post-gameplay
  Examine and describe differences in Global, Mental, Physical, and Social Health between groups using the "Patient-Reported Outcomes Measurement Information System (PROMIS)" measure described in Outcome 4. All units of measure are the same across groups. The scores will range from 2-54 with higher scores indicating better outcomes.
Semi-structured interviews with open ended questions to compare childs' and adolescents' (where appropriate), and parents' feelings about gameplay for fun, well being, quality of life in Group 1, Group 2, and Group 3 | 1 hour post-gameplay
  Using semi-structured interviews with open ended questions, we will examine and describe differences in feelings about gameplay between groups using qualitative responses gathered using semi-structured interview from Outcome 5. To be qualitatively analyzed.
Compare the parents' feelings of bonding using the "Connection & Bonding Questionnaire" with their child/adolescent in Group 1, Group 2, and Group 3 | 1 hour post-gameplay
  Examine and describe differences in feelings about parent bonding between groups using responses obtain from the "Connection & Bonding Questionnaire", a 5 item Likert-style questionnaire with responses ranging from Strongly Disagree (0) to Strongly Agree (5) and scores ranging from 0-25 with higher scores indicating a stronger connection and parent/child bond.
Compare the parents' feelings of whether the child's physical and psychological needs were met before gameplay using the "Child Needs Survey" in Group 1, Group 2, and Group 3 | 1 hour post-gameplay
  Examine and describe differences in whether the child's physical and psychological needs were met before gameplay between groups using responses from the "Child Needs Survey." A 5 item survey with 4 questions with responses of Yes, No, Unsure/Decline to Answer, and Not able/Not applicable, one visual analog-type response ranging from "Little to none" to "Fully" and one open-ended question asking parents to describe any additional needs that may or may not have been met. More "yes" answers mean a better outcome.
Compare whether the child had pain using the Visual Analog Scale in Group 1, Group 2, and Group 3 | Immediately pre-gameplay and 1 hour post-gameplay
  Examine and describe differences in whether the child had pain pre/post gameplay between groups using the Visual Analog Scales. Using a visual analog scale, have the child rate their pain pre- and immediately post-gameplay. Visual Analog Scales are a 100mm line with endpoints "none" at the 0 endpoint and "worst ever" at the 100mm endpoint. A higher score indicates a worse outcome.
Compare whether the child had stress using the Visual Analog Scale in Group 1, Group 2, and Group 3 | Immediately pre-gameplay and 1 hour post-gameplay
  Examine and describe differences in whether the child had stress pre/post gameplay between groups using the Visual Analog Scale. Using a visual analog scale, have the child rate their stress pre- and immediately post-gameplay. Visual Analog Scales are a 100mm line with endpoints "none" at the 0 endpoint and "worst ever" at the 100mm endpoint. A higher score indicates a worse outcome.
Compare whether the parent had pain using the Visual Analog Scale in Group 1, Group 2, and Group 3 | Immediately pre-gameplay and 1 hour post-gameplay
  Examine and describe differences in whether the parent had pain pre/post gameplay between groups using the Visual Analog Scale. Using a visual analog scale, have the parent rate their pain pre- and immediately post-gameplay. Visual Analog Scales are a 100mm line with endpoints "none" at the 0 endpoint and "worst ever" at the 100mm endpoint. A higher score indicates a worse outcome.
Compare whether the parent had stress using the Visual Analog Scale in Group 1, Group 2, and Group 3 | Immediately pre-gameplay and 1 hour post-gameplay
  Examine and describe differences in whether the parent had stress pre/post gameplay between groups using the Visual Analog Scale.Using a visual analog scale, have the parent rate their stress pre- and immediately post-gameplay. Visual Analog Scales are a 100mm line with endpoints "none" at the 0 endpoint and "worst ever" at the 100mm endpoint. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Thrane, PhD, RN, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data.